CLINICAL TRIAL: NCT05717608
Title: Effect Dietary Fructose on Fructose Kinetics in Type 2 Diabetes
Acronym: ERIE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Responsible Party: Principal Investigator, Max Nieuwdorp, professor, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 2022.0606 - NL82353.018.22
Record Dates: First submitted 2023-01-08; First posted 2023-02-08 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-01

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Intervention Model Description: high versus low fructose diet for 4 weeks in either caucasian or surinamese asian type 2 diabetes patients
Who Masked: Participant, Investigator
Masking Description: supplementation with either fructose or dextrose
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- high fructose in caucasian dutch type 2 diabetes subjects (Active Comparator): high (100gr/day) fructose diet for 4 weeks in type 2 diabetic subjects of Caucasian ethnicity.
  Interventions: Other: high vs low fructose in caucasian dutch or surinamese asian type 2 diabetes subjects
- low fructose in caucasian dutch type 2 diabetes subjects (Placebo Comparator): low fructose diet (<30 gram fructose intake per day isocaloric correction with dextrose) for 4 weeks in type 2 diabetic subjects of Caucasian ethnicity.
  Interventions: Other: high vs low fructose in caucasian dutch or surinamese asian type 2 diabetes subjects
- high fructose in surinamese asian type 2 diabetes (Active Comparator): high (100gr/day) fructose diet for 4 weeks in type 2 diabetic subjects of SAS ethnicity.
  Interventions: Other: high vs low fructose in caucasian dutch or surinamese asian type 2 diabetes subjects
- low fructose in surinamese asian type 2 diabetes (Placebo Comparator): low fructose diet (<30 gram fructose intake per day isocaloric correction with dextrose) for 4 weeks in type 2 diabetic subjects of SAS ethnicity.
  Interventions: Other: high vs low fructose in caucasian dutch or surinamese asian type 2 diabetes subjects

INTERVENTIONS:
Other: high vs low fructose in caucasian dutch or surinamese asian type 2 diabetes subjects — oral ingestion of food supplement for 4 weeks

SUMMARY:
Determine the kinetics of fructose metabolism and its role as a metabolic substrate following a high (100gr/day) vs low fructose diet (<30 gram fructose intake per day isocaloric correction with dextrose) in type 2 diabetic subjects of SAS or Caucasian ethnicity.

DETAILED DESCRIPTION:
The prevalence and accompanying morbidity and mortality of obesity and type 2 diabetes (T2D) is increasing on a global scale. Unfortunately the underlying (patho)physiological mechanisms are only partially understood. A key step in the development of negative health effects of metabolic disease might be via dietary fructose metabolism and its accompanying aberrant metabolite production, in which our gut microbiota plays a crucial role.

By bypassing the normal glucose metabolism pathway, fructose plays a role in the development of metabolic disease such as diabetes en fatty liver disease. The mechanism of this effect is unclear and possibly plays in the observation of ethnic specific metabolic risk factors. That is, subjects of different ethnicties (for instance South-Asian Surinamese (SAS)) have a higher risk and worse trajectory of metabolic diseases than Caucasians. Since gut microbiota is altered between these two ethnicities, we hypothesize that aberreant fructose catabolism in patients of SAS descent results in production of specific (gut microbiota derived) metabolites such as ethanol. In this study, fructose metabolism will thus be studied in patients of SAS and Caucasian Dutch descent. To this end the investigators will examine (13C stable isotope based) fructose fluxes before and after randomizing subjects into a four-week high- or low fructose diet. This study aims to elucidate the physiological and microbial catabolism of fructose and possible differences between these two ethnicities.

ELIGIBILITY:
Inclusion Criteria:

* 40 T2D patients (20 Caucasian and 20 SAS)
* 40-70 years old
* Male-female
* BMI 25-35 kg/m2
* Stable anti diabetic drugs for 3 months (metformin is obligatory)
* Stable medication use past 3 months
* Able to give informed consent

Exclusion Criteria:

* - Proton-pump inhibitor usage (known to effect gut microbiota)
* GLP1, SGLT2i or insulin use (known to effect gut microbiota)
* Antibiotic for the past 3 months (known to effect gut microbiota)
* Probiotic or symbiotic usage (known to effect gut microbiota)
* Pregnant women
* Chronic illness (including a known history of heart failure, renal failure (eGFR <30 ml/min), pulmonary disease, gastrointestinal disorders, or hematologic diseases), or other inflammatory diseases
* Active infection
* Previous intestinal (e.g., bowel resection/reconstruction) surgery
* Smoking (due to its influence on gut microbiome)
* Vegetarian diet (since they have different microbiota)
* >6 alcohol units per day or >14 alcohol units per week
* Active malignancy
* HbA1c >9% (75mmol/mol)

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-02-05 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
fructose on glucose metabolism | 4 weeks
  to correlate changes in oral fructose handling (measured by a fructose challenge test (AUC) with 13C6-labeled fructose in relation to metabolic effects on HOMA-IR and continuous glucose monitoring (Freestyle libre MAGE) at baseline and after 4 weeks of dietary intervention.

SECONDARY OUTCOMES:
changes in microbiota composition | 4 weeks
  correlate with changes in oral/fecal microbiota composition (diversity and strain)
changes in (postprandial )plasma metabolites | 4 weeks
  effects of the diet on body composition (measured via bio impedance analysis). We will also collects 24h feces and urine before each study visit to determine correlate with changes in (postprandial) untargeted plasma metabolites including endogenous ethanol

CONTACTS AND LOCATIONS:
Overall Officials: max nieuwdorp, Principal Investigator — Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Locations (1):
- Amsterdam UMC location AMC, Amsterdam, Netherlands

IPD SHARING:
Plan to Share IPD: No
not allowed due to dutch GDPR regulations